CLINICAL TRIAL: NCT03062384
Title: AT-001 for Long-term Preservation of Brain Health in Aging: The ALPHA Study
Brief Title: AT-001 for Long-term Preservation of Brain Health in Aging
Acronym: ALPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Alltech Life Sciences Inc. (Industry)
Responsible Party: Principal Investigator, Richard Ronan Murphy, M.B.B.S., Assistant Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15 0534 F6A
Record Dates: First submitted 2016-11-02; First posted 2017-02-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Oxidative Stress
Keywords: brain; health
MeSH Terms: interventions — caficrestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT-001 (Experimental): Yeast-selenium supplement
  Interventions: Dietary Supplement: AT-001
- Placebo (Placebo Comparator): Yeast supplement devoid of selenium
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AT-001
  Arms: AT-001
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if the use of a yeast-selenium supplement (AT-001) is safe in elderly subjects who do not have dementia, and further, to see if the supplement improves tests that are related to brain health.

DETAILED DESCRIPTION:
Double blind, placebo-controlled, single-center study. Approximately 40 healthy volunteers will be randomized to the study drug and 20 healthy volunteers randomized to the placebo, for a total of 60 enrolled participants.

All participants will be treated with the study drug or placebo for 12 months. Subjects will be seen in the clinic for the following visits: Screening (Day -14), Baseline (Day 0), Month 6, and End-of-Study (Month 12) while on study drug. An additional safety visit at Month 13 (four weeks after study drug discontinuation) will be required of all participants.

Participants will undergo vital signs assessment, medical history review, medication list review, and review of Adverse Events (AEs) and Serious Adverse Events (SAEs) at each visit.

Participants will undergo neuropsychological testing and routine physical examinations at the screening, baseline, and end-of-study visits.

Participants will undergo blood draws, urine collection, MRI to assess lumbar puncture safety, and lumbar puncture at the baseline and end-of-study visits.

ELIGIBILITY:
Inclusion Criteria:

* Not demented by DSM-IV criteria.
* English-speaking, to ensure compliance with cognitive testing and study visit procedures.
* Montreal Cognitive Assessment (MoCA) score at screening visit ≥24/30.
* Female participants must not be pregnant or of childbearing potential (surgically sterile or post-menopausal for >1 year).
* Stable medical condition for 3 months prior to screening visit in the opinion of the study physician.
* Non-diabetic, confirmed by fasting serum glucose <120 mg/dL and on no oral hypoglycemic agents or insulin treatment.
* No other clinically significant abnormalities on labs (CBC, chemistry panel, PT/INR, aPTT, urinalysis).
* Stable medications for 4 weeks prior to screening.
* Able to ingest oral medications.
* Physically acceptable for the study as confirmed by medial history, physical exam, neurological exam, and clinical tests in the opinion of the study physician.

Exclusion Criteria:

* Significant neurological disease, such as Parkinson's disease, brain tumor, multiple sclerosis, or seizure disorder
* Major depression in the past 12 months (DSM-IV criteria), major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse.
* History of invasive cancer within the past 2 years (excluding non-melanoma skin cancer).
* Contraindications to lumbar puncture (bleeding disorder, platelet count <100,000, anticoagulant treatment, major structural abnormality or sepsis in the area of the lumbosacral spine, or previous lower back surgery that would make LP technically difficult in the opinion of the study physician, hypersensitivity to lidocaine).
* Contraindications to MRI (pacemaker, shrapnel, metallic implants, etc).
* Clinically significant abnormalities on labs (CBC, chemistry panel, PT/INR, aPTT, urinalysis).
* Use of any investigational agents within 30 days prior to screening.
* Major surgery within eight weeks prior to the Baseline Visit.
* Severe unstable major medical illnesses, including uncontrolled cardiac conditions or heart failure (New York Heart Association Class III or IV).
* Antiretroviral therapy for human immunodeficiency virus (HIV).
* Residence in a skilled nursing facility.
* Blindness, deafness, language difficulties, or any other disability which may prevent the participant.

Excluded Medications:

* Experimental drugs.
* Coumadin, heparin, or any other anticoagulant.
* Insulin or other hypoglycemic agents.
* Supplements containing more than 50 µg selenium/day (US RDA) in the 12 weeks prior to screening.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid Aβ42 | Baseline to End-of-Study (12 months)
Serum levels of prostaglandins PGF2α and PGE2 | Baseline to End-of-Study (12 months)

SECONDARY OUTCOMES:
Urine levels of prostaglandins PGF2α and PGE2 | Baseline to End-of-Study (12 months)
Cerebrospinal fluid levels of phosphorylated and total tau protein | Baseline to End-of-Study (12 months)
Volumetric brain MRI measurements | Baseline to End-of-Study (12 months)
Neurocognitive measure: Free and Cued Selective Reminding Test (FCSRT) | Baseline to End-of-Study (12 months)
Neurocognitive measure: Trail-making test parts A and B | Baseline to End-of-Study (12 months)
Neurocognitive measure: Naming, both single letter fluency and animal naming. | Baseline to End-of-Study (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Murphy, MD, Principal Investigator — University of Kentucky; Ronan Powers, PhD, Study Director — Alltech Life Sciences Inc.; Gregory A. Jicha, MD, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky Sanders-Brown Center on Aging Clinic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No